CLINICAL TRIAL: NCT05856877
Title: Zentrale Insulinsensitivität Bei Personen Mit Typ-2-Diabetes Sowie Bei Personen Mit erhöhtem Risiko für Die Entwicklung Von Typ-2-Diabetes
Brief Title: Central Insulin Sensitivity in Individuals With Type 2 Diabetes (T2D) and at Risk for Developing T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: INCLU
Record Dates: First submitted 2023-03-21; First posted 2023-05-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Central Insulin Resistance; Diabetes Mellitus, Type 2; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal insulin spray (Active Comparator)
  Interventions: Other: Human nasal insulin
- Placebo spray (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Human nasal insulin — single dose of 160 U of human insulin as nasal spray
  Arms: Nasal insulin spray
Other: Placebo — Single dose of placebo solution as nasal spray
  Arms: Placebo spray

SUMMARY:
Beside well described peripheral effects, insulin can also affect the human central nervous system. Centrally acting insulin seems to have an influence e.g. on whole-body metabolism and food intake. Targeting insulin receptors in the central nervous system can modulate peripheral insulin sensitivity as well as pancreatic insulin secretion. In humans, the effect of insulin can be measured in different brain areas as estimate of central nervous insulin sensitivity. Reduced central nervous insulin sensitivity, called "central insulin resistance," has been associated, for example, with obesity, unfavorable body fat distribution, and impaired cognitive functionality. Recently novel subtypes and risk clusters of diabetes and prediabetes have been identified. In this study the investigators want to investigate and compare central nervous insulin sensitivity as well as cognitive function in the different diabetes and prediabetes risk clusters.

ELIGIBILITY:
Inclusion Criteria:

1. manifest diabetes mellitus type 2 with initial diagnosis ≤ 10 years ago, defined as

   * a fasting blood glucose greater than 126 mg/dl and/or
   * a blood glucose greater than 200 mg/dl at the 120 minute time point in the oral glucose tolerance test with 75 g glucose and/or
   * an HbA1c greater than 6.5%
2. or a currently existing increased risk of developing type 2 diabetes, defined as

   * prediabetes, defined as

     * elevated fasting blood glucose (IFG), fasting blood glucose between 100 and 125 mg/dl) and/or
     * impaired glucose tolerance (IGT), 120-minute oral glucose tolerance test blood glucose between 140 and 199 mg/dl) and/or
     * HbA1c between 5.7% and 6.4% with
   * and/or at least one of the following factors indicating an increased risk for developing type 2 diabetes mellitus:

     * previously existing prediabetes and/or
     * recent-onset gestational diabetes, and/or
     * positive family history (1st degree family members) for type 2 diabetes mellitus and/or
     * BMI greater than 27 kg/m2
3. or no manifest diabetes mellitus type 2 and no currently existing increased risk for developing type 2 diabetes (control group: BMI 18.5 to 24.5 kg/m2)
4. female and male (1:1), voluntary adults
5. at least 18 years old and able to give consent
6. understanding of study explanations and instructions
7. consent to information in case of unexpected proven pathological findings.

Exclusion Criteria:

* Only in subjects without manifest diabetes mellitus type 2: Taking medications that affect sugar metabolism (e.g., antidiabetic medications or glucocorticoids).
* Diabetes mellitus type 1 or Latent autoimmune diabetes in the adult (GAD and/or IA2 antibodies positive)
* MODY (Maturity onset Diabetes of the Young)
* Decompensated diabetes mellitus type 2 (HbA1c greater than 9.6% and/or fasting blood glucose > 230 mg/dl)
* BMI < 18.5 or > 45 kg/m2
* Individuals wearing non-removable metal devices in or on the body such as:

  * pacemakers
  * artificial heart valves
  * metal prostheses
  * implanted magnetic metal parts (screws, plates from surgery)
  * coils
  * metal splinters/garnet chips
  * fixed braces
  * retainers going over more than four teeth
  * acupuncture needle
  * Insulin pump
  * intraport
  * Tattoos, eye shadow, etc.
* there is a pregnancy or pregnancy cannot be excluded
* breastfeeding women
* Individuals with impaired temperature sensation and/or increased sensitivity to heating of the body.
* symptomatic coronary heart disease, heart failure greater than NYHA 3, previous heart attack
* Condition following stroke
* Individuals with hearing disease or increased sensitivity to loud sounds
* Persons with claustrophobia (fear of place)
* Minors or subjects incapable of giving consent
* Subjects who have had an operation less than 3 months ago
* Acute illness or infection within the last 4 weeks
* Severe neurological or psychiatric diseases, e.g. severe depression (at least 29 points according to BDI II), schizophrenia or bipolar disorder.
* Use of centrally acting drugs
* Known presence of malignant disease within the last 5 years
* Diseases of the pancreas
* Systemic infection (CRP > 1 mg/dl)
* Following bariatric surgery
* Antibiotic therapy within the last 4 weeks prior to study inclusion
* No consent to be informed about incidentally discovered pathological findings
* Participation in interventional trials and receipt of investigational medication in the last 30 days
* Severe diabetic complications such as chronic kidney disease (KDIGO CKD greater than G4) or severe proliferative retinopathy
* Subjects with hemoglobin levels Hb<10.5g/dl (for women), Hb<11.5g/dl (for men)
* Other medical conditions that, in the opinion of an investigator, may jeopardize the success of the study or indicate that the subject may be at risk of harm
* Allergic diseases to any of the substances used

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of brain insulin sensitivity in different age, weight, sex and metabolic risk groups | 30 minutes after Administration of nasal insulin
  fMRI measurement will be performed before and after administration of 160 U human insulin or placebo as nasal spray. Changes in regional brain activity will be quantified by cerebral blood flow and blood oxygenation dependent (BOLD) signal to assess regional brain insulin sensitivity. Brain insulin sensitivity will be compared between 5 groups (T2DM-high risk group, T2DM-low risk group, elevated risk for developing T2DM-high risk group, elevated risk for developing T2DM-low risk group, lean and healthy group). Persons are categorized into normal weight and overweight/obese based on the Body Mass Index (BMI). Age groups are build based on a median split. Metabolic risk groups are build based on Ahlqvist-criteria (T2DM) and based on Wagner-criteria (elevated risk for developing T2DM).
Comparison of cognitive function between subtype clusters of different metabolic groups (increased risk for developing manifest type 2 diabetes cluster, manifest type 2 diabetes cluster) | 45 minutes
  CANTAB test will be performed
Comparison of the blood-brain-barrier permeability in different age, weight, sex and metabolic risk groups | 30 minutes after Administration of nasal insulin
  fMRI measurement will be performed before and after administration of 160 U human insulin or placebo as nasal spray. Changes in blood-brain-barrier permeability will be quantified by cerebral blood flow and blood oxygenation dependent (BOLD) signal to assess blood-brain-barrier permeability. blood-brain-barrier permeability will be compared between 5 groups (T2DM-high risk group, T2DM-low risk group, elevated risk for developing T2DM-high risk group, elevated risk for developing T2DM-low risk group, lean and healthy group). Persons are categorized into normal weight and overweight/obese based on the Body Mass Index (BMI). Age groups are build based on a median split. Metabolic risk groups are build based on Ahlqvist-criteria (T2DM) and based on Wagner-criteria (elevated risk for developing T2DM).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Germany